CLINICAL TRIAL: NCT06283576
Title: Pancreatic Cancer Initial Detection Via Liquid Biopsy
Acronym: PANCAID
Status: Enrolling by invitation | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Matthias Löhr, Professor of Gastroenterology & Hepatology, Karolinska University Hospital
Other Study IDs: PANCAID-00-08
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer; IPMN, Pancreatic; Individuals at Risk; Chronic Pancreatitis
Keywords: diabetes mellitus; smoking
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Intraductal Neoplasms; Pancreatitis, Chronic; Diabetes Mellitus; Smoking | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liquid biopsy: ct-DNA, extracellular vesicles, proeomics, metabolomics, CTC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pancreatic cancer, early: Early pancreatic cancer, T1/T2 NoM0
  Interventions: Diagnostic Test: Liquid biopsy
- IPMN
  Interventions: Diagnostic Test: Liquid biopsy
- Pancreatic cancer, advanced: Advance pancreatic cancer T1-4, Nx, Mx
  Interventions: Diagnostic Test: Liquid biopsy
- Healthy controls
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — Blood will be drawn upon clinical diagnosis / prior to biopsy/surgical resection for "ground truth"

SUMMARY:
The overall rationale of PANCAID is to provide a diagnostic blood test for early diagnosis of pancreatic cancer. With a set of different liquid biopsy methods, it is the aim to measure these markers in well-defined patient cohorts. For the entire series of these studies, the following groups are planned: 1) Histologically proven early-stage pancreatic cancer (e.g. T1a/b and T2 carcinomas [N0M0]); 2) Intraductal papillary mucinous neoplasia (IPMN) that were operated with verification of the benign, premalignant or malignant histology; 3) ordinary branched-duct IPMN; 4) individuals at risk (IAR) with and without IPMN, with and without known hereditary cancer gene (e.g. BRCA2); 5) a high risk group of patients with chronic pancreatitis, aged 55-65, who are heavy smokers (≥40 PY), with newly onset diabetes mellitus (NODM).

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of or elevated risk for pancreatic ductal adenocarcinoma (PDAC); intraductal papillary mucinous neoplasias (IPMN); individuals at risk (IAR) for pancreatic cancer

Exclusion Criteria:

* other malignant condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults capable of giving informed consent to give blood for liquid biopsy coming to the University Hospitals of Stockhol (Karolinska) and Umeå
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer detection | Up to 4 weeks after surgery
  Liquid biopsy test(s) detecting pancreatic cancer on biobanked, archival samples of patients with histologically confirmed pancreatic lesions (PDAC, IPMN, pancreatitis).

SECONDARY OUTCOMES:
Overall survival | 1 month - 24 months after surgical resection of the tumor
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrocentrum, KarolinskaUniversity Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request to the PANCAID consortium
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completion of the study
Access Criteria: Clearance from Scientifc and Ethical Advisory Board of PANCAID (see www.pancaid-project.eu/)
URL: http://www.pancaid-project.eu/